CLINICAL TRIAL: NCT02924805
Title: Telemedical Versus Conventional Emergency Care of Hypertensive Emergencies and Urgencies
Brief Title: Telemedical Versus Conventional Emergency Care of Hypertensive Emergencies
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: TECH
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Hypertensive Emergency; Hypertensive Urgency
MeSH Terms: conditions — Hypertensive Crisis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Telemedicine group: Cases of hypertensive emergencies and urgencies in which the prehospital emergency care was performed by on-scene paramedics, guided by a qualified physician in a teleconsultation center.
  Interventions: Other: Telemedical care
- Control group: Historical cases of of hypertensive emergencies and urgencies in which the prehospital emergency care was carried out by on-scene emergency medical service physicians (conventional care).

INTERVENTIONS:
Other: Telemedical care — Telemedically guided care based on a standard operating procedure
  Groups: Telemedicine group

SUMMARY:
Comparison of telemedical prehospital emergency care and conventional on-scene physician based care of hypertensive emergencies and urgencies. The adherence to current Guidelines should be researched.

DETAILED DESCRIPTION:
Telemedically guided cases of hypertensive emergencies (april 2014 - March 2015) and urgencies are compared with a historical control group of conventional emergency medical service physician care on-scene for these scenarios. The historical control group is a time period prior to implementation of the telemedicine system and after a research project with a precursor telemedicine system. No telemedical support but only conventional on-scene EMS physician care was available (November 2013 - March 2014).

ELIGIBILITY:
Inclusion Criteria:

* prehospital diagnosis of hypertensive emergency of hypertensive urgency

Exclusion Criteria:

Prehospital diagnoses of:

* pulmonary edema
* aortic dissection
* acute coronary syndrome
* acute stroke
* acute respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whith a prehospital diagnosis of hypertensive emergency or urgency
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure difference between initial contact and emergency room handover | 2 hours

SECONDARY OUTCOMES:
Difference of heart rate between initial contact and emergency room handover | 2 hours
Magnitude of blood pressure reduction using categories | 2 hours
  To measure guideline adherence blood pressure (BP) reductions were evaluated with four categories: no BP reduction, reduction <= 25%, reduction >25-30%, reduction > 30% (BP difference between initial contact and emergency room handover)

OTHER OUTCOMES:
Analysis of administered antihypertensive agents | 2 hours
context specific quality of medical history and documentation | 2 hours
  Analysis of medical history and vital parameter documentation completeness

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Ch Brokmann, Dr. med., Principal Investigator — University Hospital Aachen, Germany
Locations (1):
- University Hospital Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No